CLINICAL TRIAL: NCT02441751
Title: Intraoperative Repolarisation - Etiology and Relevance for the Decision Making by Anesthesiologists in the Management of Volume Substitution and Transfusion
Brief Title: Intraoperative Volume Management and QT Interval
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: EK110032015
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Blood Loss, Surgical
Keywords: Electrocardiography; Hemorrhage; Monitoring, Intraoperative
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- bleeding: intraoperative blood loss > 500 ml
  Interventions: Procedure: intra-operative blood loss
- no bleeding: intraoperative blood loss < 500 ml

INTERVENTIONS:
Procedure: intra-operative blood loss — surgery in the urology and orthopedics
  Groups: bleeding

SUMMARY:
QT interval changes is measured during all phases of the operation. The protocol is focusing at intraoperative bleeding events and is also observing QT interval changes during anesthetic and operative procedures.

DETAILED DESCRIPTION:
Prolongation of the QT interval is associated with functional torsade de points, re-entry, and sudden death (see reference). Variations of QT-interval caused by changes in the volume status of the patient during an operation remained unclear. QT interval changes will be monitored during the surgery with the focus of the influence of sudden blood loss, volume substitution by crystalloids, blood and blood products. The effect of surgical procedures on the QT-interval (e.g. clamping of kidney artery) will be observed as well as the association of intra-operative QT-interval alterations with postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification 2 - 3
* patients after consent

Exclusion Criteria:

* Children,
* pregnant women,
* patients not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients for major surgery in urology and orthopedics
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change in QT-time | during operation

SECONDARY OUTCOMES:
postoperative incidents/disturbance rhythm of the heart | 2 days
  association to intraoperative repolarisation-disturbance / QT-prolongation
survival | 1 year
  association to intraoperative repolarisation-disturbance / QT-prolongation

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Richter, M.D., Study Director — University Hospital Dresden, TU Dresden
Locations (1):
- Dept. of Anesthesia and Intensive Care, University Hospital, Technische Universität Dresden, Dresden, Germany

REFERENCES:
- [Background] Straus SM, Kors JA, De Bruin ML, van der Hooft CS, Hofman A, Heeringa J, Deckers JW, Kingma JH, Sturkenboom MC, Stricker BH, Witteman JC. Prolonged QTc interval and risk of sudden cardiac death in a population of older adults. J Am Coll Cardiol. 2006 Jan 17;47(2):362-7. doi: 10.1016/j.jacc.2005.08.067. PMID 16412861